CLINICAL TRIAL: NCT05273294
Title: Ultrasound Measurements of Circular Cartilage Transverse Diameter Were Used for the Selection of Surgical Tracheal Catheter in Younger Children
Brief Title: Ultrasound Measurements of Circular Cartilage Transverse Diameter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ultrasound measurements
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Ultrasound Therapy; Complications; Transverse Diameter of Cricoid Cartilage; Endotracheal Intubation; Children

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): Anesthesiologist will convenient color ultrasound high frequency 12MHZ array probe perpendicular to the neck, by the glottal down, until the thyroid isthmus, and ring cartilage level, ring cartilage level diameter by ultrasound, to avoid the effect of inspiration and breath on airway diameter, measurement timing should choose after anesthesia induction, mask pressure gas 1min, suspended pressure ventilation for 5s, ultrasonic measurement time is not more than 10s.Repeated measurements were averaged three times, and the maximum outer diameter of the catheter was selected, that is, the maximum outer diameter was selected closest to the measured value.
  Interventions: Device: Portable color Doppler ultrasound system
- Control group (No Intervention): tracheal catheter models are usually selected through traditional experience, according to the age formula in Clinical Anesthesiology, People's Health Press (i. e., 2.5 for preterm infants, 3.5 at 1-6 months, 4.0 at 6-12 months).

INTERVENTIONS:
Device: Portable color Doppler ultrasound system — In the ultrasound group, the catheter type was selected according to the results of ultrasonic measurement of transverse diameter of cricoid cartilage after induction of general anesthesia, and tracheal intubation was performed with ordinary laryngoscope after measurement
  Arms: Ultrasound group

SUMMARY:
This study with children under 1 age of elective surgery as the research subjects, according to the cross diameter, compared with the traditional method of empirical catheter model, analyze the success rate, completion time of intubation, endotracheal intubation attempts and complications, explore the clinical value of pediatric endotracheal technology, to provide new ideas and methods for clinical practice.

DETAILED DESCRIPTION:
A total of 90 children younger than 1 year old who underwent endotracheal intubation under elective general anesthesia in Shengjing Hospital affiliated to China Medical University from January 2022 to June 2022.Ninety patients were randomized by placing the numbers of the experimental and control patients in opaque envelopes in patient order.After having the envelope sealed and scrambled, number it in the order of 1 to 2.When each new patient entered the study, an envelope was opened and entered according to the allocation protocol in the envelope.The procedure was repeated for the patients in each group.The Informed consent was signed by an uninformed anesthesia assistant, and all patients included in the experiment and their families were unaware of the grouping.Of these, 47 were male, 43 females, ASA grade I or II, age less than 1 year, height (63.6±9.13) cm, and weight (7.55±7.37) kg.

All children with routine preoperative fasting, postoperative monitoring monitoring electrocardiogram (ECG), blood pressure (BP) and blood oxygen saturation (SPO2), mask oxygen inhalation, maintain SPO298%, intravenous induction, intravenous sufentanil 2ug/kg, Etomidate 0.2mg/kg, rouronium 0.6mg/kg, manually assisted ventilation until muscle release completely started.Ultrasonic measurement group, the anesthesiologist, who was trained by professional physician and not know the study plan, will probe ultrasonic probe with coupling agent after long axis with the neck on the sternoclavicular articulation point 0.5 cm place to get the cricoOD cartilage parallel plane image, obtain patients expiratory pause at the end of the clearance of cricoOD cartilage ring diameter image, the average value was taken after obtaining repeated measurements 3 times. Select the tracheal duct model based on the measured transverse diameter of circular cartilage, That is, the largest tracheal tube with an outer diameter smaller than the transverse diameter of the circular cartilage, Perform tracheal intubation, Determine whether the catheter model is suitable according to the air leakage test.Air leakage test: the sleeve is not inflated, adjust the oxygen flow of the anesthesia machine by 3.0 L/min, adjust the pressure preset of the APL valve, if the pressure of the APL valve is set to 10cm H2O; if the pressure of the APL valve is set to 20cm H2O, the diameter is too large to be clinically suitable in between.Double lung ausculatory respiratory sound symmetry to determine intubation depth, adjust depth for post-fixation catheter, mechanical ventilation, pressure control ventilation mode, pressure of 10-20cm H2O, respiratory of 22-24 beats/min, adjusted to intraoperative PetCO2 levels to maintain it at 35-45mmHg.The measurement of circular cartilage transverse diameter, tracheal intubation operation and anesthesia management operation of the above children were completed by two skilled anesthesiologists, and the data were recorded.Radial and internal jugular vein puncture was performed, and immediate arterial pressure and central venous pressure were measured.

Selection of tracheal catheter type:

Ultrasound group: anesthesiologist will convenient color ultrasound high frequency 12MHZ array probe perpendicular to the neck, by the glottal down, until the thyroid isthmus, and ring cartilage level, ring cartilage level diameter by ultrasound, to avoid the effect of inspiration and breath on airway diameter, measurement timing should choose after anesthesia induction, mask pressure gas 1min, suspended pressure ventilation for 5s, ultrasonic measurement time is not more than 10s.Repeated measurements were averaged three times, and the maximum outer diameter of the catheter was selected, that is, the maximum outer diameter was selected closest to the measured value.The outer diameter of the endotracheal catheter used in Shengjing Hospital, China Medical University is shown in Table 4.

Control group: tracheal catheter models are usually selected through traditional experience, according to the age formula in Clinical Anesthesiology, People's Health Press (i. e., 2.5 for preterm infants, 3.5 at 1-6 months, 4.0 at 6-12 months).

Observation and record index:

The success rate of complete intubation, the time required for endotracheal intubation, the number of tracheal intubation attempts, and the complications were recorded.Statistical analysis was conducted between the transverse diameter, age, height and weight and the outer diameter (The outer diameter, OD).The time of tracheal intubation in this study was calculated from the completion of oxygen inhalation immediately after the insertion into the laryngeal lens to the successful insertion of the appropriate tracheal catheter.

ELIGIBILITY:
Inclusion Criteria:

* Children under 1 year old who received selective general anesthesia for endotracheal intubation in Shengjing Hospital affiliated to China Medical University.

Exclusion Criteria:

* Previous history of difficult intubation, or a history of anesthesia-related adverse events.
* There are respiratory anatomical abnormalities, such as cleft lip and palate, throat stenosis, etc
* There are temporomandibular joint lesions, maxillofacial scar contracture, small jaw, etc.
* Limited head and neck activity, such as neck scar contracture, excessive obese neck shortening, cervical trauma or lesion, cervical huge tumor, congenital torticollis, etc.
* There are acute and chronic respiratory diseases, such as respiratory tract infection and bronchial asthma.
* There are diseases affecting laryngeal exposure, such as tonsil hypertrophy, tongue hypertrophy, vocal coral polyps, laryngeal edema.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of endotracheal intubation | 24 hours after surgery
  The single success rate of endotracheal intubation between the two groups
The during time of tracheal intubation | 24 hours after surgery
  Time required for endotracheal intubation

SECONDARY OUTCOMES:
Complications of endotracheal intubation | 24 hours after surgery
  Tracheal intubation-related complications were recorded within 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yanchao Yang, PHD, Principal Investigator — Shengjing Hospital
Locations (1):
- Junchao Zhu, Shenyang, China